CLINICAL TRIAL: NCT01988194
Title: Pragmatic Randomized Controlled Trial of Adjunct Acupuncture vs Usual Care Among Hospitalized Patients
Brief Title: Pragmatic Research eXamining Inpatient Symptoms
Acronym: PRAXIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13-11353
Record Dates: First submitted 2013-11-05; First posted 2013-11-20 (Estimated); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Postoperative Pain; Nausea; Vomiting; Anxiety; Depression
Keywords: acupuncture; postoperative pain; nausea; vomiting; anxiety; depression; hospitalization; inpatient
MeSH Terms: conditions — Pain, Postoperative; Nausea; Vomiting; Anxiety Disorders; Depression | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual care (No Intervention): Participants will receive usual care in the hospital.
- Usual care with acupuncture (Experimental): Participants will receive usual care with acupuncture treatments up to four days per week for the duration of their hospital stay.
  Interventions: Procedure: Acupuncture

INTERVENTIONS:
Procedure: Acupuncture — Acupuncture treatments will be provided in patient rooms up to four days per week for the duration of their hospital stay. Treatments will be consistent with how acupuncture is typically practiced: acupuncturists will diagnosis patients according to principles of traditional Chinese medicine (TCM); and treatments will be individualized to the patients. Duration of assessment, needle placement and retention will be 20-30 minutes.
  Arms: Usual care with acupuncture

SUMMARY:
Many hospitalized patients experience pain during their hospital stay, and less than half report adequate pain relief. Common treatments for pain include opioid medications, which have associated side effects and complications. Research has shown that acupuncture is effective for surgical, postoperative and cancer-related pain, nausea, and vomiting. More research is needed on the effectiveness of adding acupuncture to routine care for hospitalized patients. The objective of this study is to examine the effectiveness of acupuncture delivered in a "real-world" setting according to the principles of traditional Chinese medicine among hospitalized patients to manage pain and other symptoms. 250 hospitalized participants will be randomized in a 1 to 1 ratio to receive either 1) usual care or 2) usual care with acupuncture offered (125 in each group). The primary outcome measure will be change in daily pain intensity. Data on other symptoms, such as nausea, vomiting, anxiety, and depression, as well as functionality and quality of life will be collected in person, on a web-based survey, or via telephone follow-up. The aims of the study are to examine the effectiveness of acupuncture to manage pain and other symptoms among hospitalized patients; to evaluate the impact of acupuncture on patient satisfaction among hospitalized patients; and to estimate costs and cost-effectiveness of acupuncture among a subset of hospitalized patients.

The investigators hypothesize that compared to hospitalized patients receiving usual care alone, hospitalized patients receiving acupuncture will have:

1. decreased pain severity
2. higher patient satisfaction

ELIGIBILITY:
Inclusion Criteria:

* English or Spanish speaking
* Admitted to Mt Zion Hospital for a minimum anticipated length of stay for at least 4 days
* Aged 18 or older
* In a ward included in the roll out of the Osher Center's acupuncture program at Mt Zion

Exclusion Criteria:

* Unstable medical condition (e.g., severe pulmonary disease, myocardial infarction, severe depression, patients in the intensive care unit)
* Acupuncture contraindication (e.g., sepsis, endocarditis)
* Inability to consent or complete surveys (e.g., cognitive or communication impairment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Self-reported pain | Participants will be followed for the duration of hospital stay, an expected average of 6 days
  Daily pain intensity will be measured on a 0-10 numeric rating scale. The APS Patient Outcome Questionnaire will also be administered each day to measure pain severity and relief; impact of pain on activity, sleep, and negative emotions; side effects of treatment; helpfulness of information about pain treatment; and ability to participate in pain treatment decisions.

SECONDARY OUTCOMES:
Self-reported nausea and vomiting | Participants will be followed for the duration of hospital stay, an expected average of 6 days
  Daily nausea and vomiting symptoms will be measured using the 2-question Postoperative Nausea and Vomiting Scale.
Self-reported anxiety and depression | Participants will be followed for the duration of hospital stay, an expected average of 6 days
  Every other day, anxiety and depression will be measured using the 30-item Profile of Mood States questionnaire.
Functionality and quality of life | Participants will be followed for the duration of hospital stay and for several days after hospital discharge, an expected total average of 9 days
  Functionality and quality of life will be measured using the EQ-5D questionnaire at baseline and within 3 days of hospital discharge.
Patient satisfaction | Participants will be followed for the duration of hospital stay and for several days after hospital discharge, an expected total average of 9 days
  Within 3 days after hospital discharge, participants will be contacted to answer questions about their recent hospital stay, including questions about communication with clinicians, responsiveness of hospital staff, cleanliness and quietness of the hospital environment, pain management, and overall experience in the hospital.
Self-reported global well-being | Participants will be followed for the duration of hospital stay, an expected average of 6 days
  Every other day, global well-being will be measured using the single item Arizona Integrated Outcomes Scale.
Self-reported global rating of change | Participants will be followed for the duration of hospital stay, an expected average of 6 days
  On the last day of hospitalization, the patient's minimal clinically important difference in pain will be measured using the single item Patient Global Impression of Change Scale.

OTHER OUTCOMES:
Hospital costs and charges | Participants will be followed for the duration of hospital stay, an expected average of 6 days
  After discharge from the hospital, data from the medical record will be extracted to determine the diagnosis group, length of stay, and costs of medications used for pain, anxiety, nausea/vomiting, and anesthesia.
Use of medications | Participants will be followed for the duration of hospital stay, an expected average of 6 days
  Data about medication use will be extracted from the participant's medical chart, including type(s) of analgesics, total dose, the number of agents, whether opioids and/or adjuncts were required, and mode of delivery.
Time to ambulation | Participants will be followed for the duration of hospital stay, an expected average of 6 days
  Data will be extracted from the participant's medical chart to determine date of ambulation.
30 day readmission | Participants will be followed for the duration of hospital stay and for up to 30 days after hospital discharge, for a total expected average of 36 days
  Data will be extracted from the participant's medical chart to determine whether the participant has been readmitted to the hospital within 30 days of discharge.
Length of hospital stay | Participants will be followed for the duration of hospital stay, an expected average of 6 days
  Data will be extracted from the participant's medical chart to determine length of hospital stay.
Foley catheter removal | Participants will be followed for the duration of hospital stay, an expected average of 6 days
  Data will be extracted from the participant's medical chart to determine date of Foley catheter removal.

CONTACTS AND LOCATIONS:
Overall Officials: Maria T Chao, DrPH, MPA, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Medical Center at Mount Zion, San Francisco, California, United States

REFERENCES:
- [Background] Dix P, Sandhar B, Murdoch J, MacIntyre PA. Pain on medical wards in a district general hospital. Br J Anaesth. 2004 Feb;92(2):235-7. doi: 10.1093/bja/aeh052. PMID 14722175
- [Background] Apfelbaum JL, Chen C, Mehta SS, Gan TJ. Postoperative pain experience: results from a national survey suggest postoperative pain continues to be undermanaged. Anesth Analg. 2003 Aug;97(2):534-540. doi: 10.1213/01.ANE.0000068822.10113.9E. PMID 12873949
- [Background] Conway Morris A, Howie N. Pain in medical inpatients: an under-recognised problem? J R Coll Physicians Edinb. 2009 Dec;39(4):292-5. doi: 10.4997/JRCPE.2009.401. PMID 21152463
- [Background] Whelan CT, Jin L, Meltzer D. Pain and satisfaction with pain control in hospitalized medical patients: no such thing as low risk. Arch Intern Med. 2004 Jan 26;164(2):175-80. doi: 10.1001/archinte.164.2.175. PMID 14744841
- [Background] Benyamin R, Trescot AM, Datta S, Buenaventura R, Adlaka R, Sehgal N, Glaser SE, Vallejo R. Opioid complications and side effects. Pain Physician. 2008 Mar;11(2 Suppl):S105-20. PMID 18443635
- [Background] Sun Y, Gan TJ, Dubose JW, Habib AS. Acupuncture and related techniques for postoperative pain: a systematic review of randomized controlled trials. Br J Anaesth. 2008 Aug;101(2):151-60. doi: 10.1093/bja/aen146. Epub 2008 Jun 2. PMID 18522936
- [Background] Ezzo JM, Richardson MA, Vickers A, Allen C, Dibble SL, Issell BF, Lao L, Pearl M, Ramirez G, Roscoe J, Shen J, Shivnan JC, Streitberger K, Treish I, Zhang G. Acupuncture-point stimulation for chemotherapy-induced nausea or vomiting. Cochrane Database Syst Rev. 2006 Apr 19;(2):CD002285. doi: 10.1002/14651858.CD002285.pub2. PMID 16625560
- [Background] Lee A, Fan LT. Stimulation of the wrist acupuncture point P6 for preventing postoperative nausea and vomiting. Cochrane Database Syst Rev. 2009 Apr 15;(2):CD003281. doi: 10.1002/14651858.CD003281.pub3. PMID 19370583
- [Derived] Chao MT, Chang A, Reddy S, Harrison JD, Acquah J, Toveg M, Santana T, Hecht FM. Adjunctive acupuncture for pain and symptom management in the inpatient setting: protocol for a pilot hybrid effectiveness-implementation study. J Integr Med. 2016 May;14(3):228-38. doi: 10.1016/S2095-4964(16)60252-2. PMID 27181130